CLINICAL TRIAL: NCT05449756
Title: A Virtual, Decentralised Observational Follow-up Study Investigating Feeding Patterns in Infancy and the Associated Parent-reported Allergic Manifestations, Allergies and Infections in Childhood.
Brief Title: A Follow-up Study With Children Who Participated in the TEMPO Study in Their First Year of Life
Status: Recruiting | Type: Observational
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: EBB18TA23570
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Allergy; Infections
MeSH Terms: conditions — Hypersensitivity; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children who participated in randomised clinical trail, called TEMPO, in their first year of life: Children who participated in randomised clinical trail, called TEMPO, in their first year of life
  Interventions: Other: Self-administered questionnaires

INTERVENTIONS:
Other: Self-administered questionnaires — Three-monthly self-administered digital questionnaires (accessed on smartphone, tablet or computer)

SUMMARY:
This is a follow-up study of a randomised clinical trial, called TEMPO (a double-blind randomized clinical trial investigating infant formula and human breast milk consumption), in which infants participated in their first year of life. The investigators like to know if these children develop allergies or infections in childhood and whether their feeding pattern in infancy plays a role.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to participate in the TEMPO Follow-Up study in case:
* they completed the final (12 months) visit in the TEMPO study.
* parents agree that their contact details will be shared with a third party for study purposes.
* parents agree that data collected in the TEMPO study will be used in the TEMPO Follow-Up study.
* parents provide written informed consent for participation in the TEMPO Follow-Up in accordance with local law.

Exclusion Criteria:

* Parents who do not have a smartphone, tablet or personal computer with internet access.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: TEMPO study subjects who completed the final (12 months) visit in the TEMPO study and consented to be approached for follow-up
Sampling Method: Non-Probability Sample
Enrollment: 705 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Parent-reported symptoms of allergies and infections | 7.5 years
  The occurrence of parent-reported - symptoms suggestive of allergies and infections
Parent-reported use of medications and/or a medical device | 7.5 years
  The occurrence of parent-reported - use of medications and/or a medical device to prevent or relieve symptoms suggestive of allergies and infections
Parent-reported - hospitalisations and visits to the emergency room | 7.5 years
  The occurrence of parent-reported - hospitalisations and visits to the emergency room for symptoms suggestive of allergies and infections

CONTACTS AND LOCATIONS:
Locations (1):
- PreCare Trial & Recruitment, Beek, Netherlands

IPD SHARING:
Plan to Share IPD: No